CLINICAL TRIAL: NCT02445924
Title: Micro RNA Genetic Signature in Non-small Cell Lung Cancer Egyptian Patients
Brief Title: Micro RNA Genetic Signature in NSCLC Egyptian Patients
Status: Completed | Type: Observational
Sponsor: Adel Salah Bediwy (Other)
Responsible Party: Sponsor-Investigator, Adel Salah Bediwy, Assistant Professor of Chest Diseases, Faculty of Medicine, Tanta University
Organization: Tanta University (Other)
Other Study IDs: 2858/11/14
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: genetic signature; non-small cell lung cancer; micro RNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, bronchial lavage, bronchial biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control group 1: ten non smoker volunteers
- Control group 2: ten smoker volunteers
- NSCLC patients: twenty NSCLC patients confirmed by pathological examination of bronchoalveolar examination (BAL), brush and/or biopsy

SUMMARY:
This study will be carried out on 40 subjects at Chest department Tanta university hospital

The subjects will be classified into three groups:

* Group I: will include ten non smoker volunteers (control group I).
* GroupII: will include ten smoker volunteers (control groupII).
* Group III: will include twenty NSCLC patients confirmed by pathological examination of bronchoalveolar examination (BAL), brush and/or biopsy.

DETAILED DESCRIPTION:
The patients and control groups will be subjected to the following:

* Complete history taking and complete general examination.
* Complete chest examination.
* Radiological assessment including chest x ray (posteroanterior and lateral view).
* Computed tomography (CT) chest for all patients in group III and when needed in group I and II.
* Laboratory investigations:

  * Complete blood picture
  * Fasting and post parandial blood sugar level
  * liver function tests
  * kidney function tests (urea and creatinine).
  * Prothrombine time and activity.
  * Zeil-Neelsen staining of sputum.
  * Tumour markers including α Fetoprotein, Carcino Embryonic antigen (CEA), CA19-9, CA 125, CA15-3 and others.
* Venous blood samples will be collected from peripheral blood (5 ml) under complete aseptic technique. Serum samples will be obtained by centrifugation. Isolation of total RNA from serum pools will be performed. RNA profiles and quantification will be assessed using Microarray.
* Lung biopsy either transbronchial via bronchoscopy or peripherally via ultrasound , CT guided, thoracoscopy or open lung biopsy will be performed with isolation of total RNA from lung tissue biopsy. RNA profiles and quantification will be assessed using Microarray.
* Bronchoalveolar lavage will be performed with isolation of total RNA from it. RNA profiles will be assessed using Microarray.

Ethical considerations:

1. Informed consent will be taken from all subject's and include:

   A. The aim of research. B. All data are confidential. C. All data will be used in research only.
2. For patient's privacy:

   A. There will be a code number for each patient in special folder. B. The results of research will be used in scientific publishing only.
3. Unexpected risks that appear during the courses of research will be cleared to the participants and the ethical committee on time.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients:

Non small cell lung cancer patients recently diagnosed who did not receive chemotherapy, surgery or radiation therapy.

-

Exclusion Criteria:

* Exclusion criteria for patients:
* Diagnosis of asthma or COPD.
* Broncheiactasis.
* upper/lower respiratory tract infection in the preceding 4 weeks.
* Active pulmonary tuberculosis.
* Associated cancer beside lung cancer.
* Patients who received chemotherapy, surgery or radiation therapy previous to the sample collection.

Exclusion criteria for control subjects:

* Diagnosis of asthma or COPD.
* Broncheiactasis.
* Upper/lower respiratory tract infection in the preceding 4 weeks.
* Active pulmonary tuberculosis
* Smoking in group I.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be carried out on 40 subjects at Chest department Tanta university hospital.
  The subjects will be classified into three groups:
  * Group I: will include ten non smoker volunteers (control group I).
  * GroupII: will include ten smoker volunteers (control groupII).
  * Group III: will include twenty NSCLC patients confirmed by pathological examination of bronchoalveolar examination (BAL), brush and/or biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Detect micro RNA genetic signature pattern in non-small cell lung cancer Egyptian patients assessed using Microarray | one year

CONTACTS AND LOCATIONS:
Overall Officials: Amgad A Farahat, MD, Study Chair — Chest Department, Faculty of Medicine, Tanta University; Ayman H Abd El-Zaher, MD, Principal Investigator — Chest Department, Faculty of Medicine, Tanta University; Said M Hammad, MD, Principal Investigator — Clinical Pathology Department, Faculty of Medicine, Tanta University; Adel S Bediwy, MD, Principal Investigator — Chest Department, Faculty of Medicine, Tanta University; Ayman A Al Saka, MD, Principal Investigator — Pathology Department, Faculty of Medicine, Tanta University; Samar A Mansour, Master, Principal Investigator — Chest Department, Faculty of Medicine, Tanta University; Abdel-Aziz A Zidan, PHD, Principal Investigator — Director of Genomics and Proteomics Unit, Center of Excellence in Cancer Research, Tanta University
Locations (1):
- Chest Department, Faculty of Medicine, Tanta University, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Background] Tang D, Shen Y, Wang M, Yang R, Wang Z, Sui A, Jiao W, Wang Y. Identification of plasma microRNAs as novel noninvasive biomarkers for early detection of lung cancer. Eur J Cancer Prev. 2013 Nov;22(6):540-8. doi: 10.1097/CEJ.0b013e32835f3be9. PMID 23462458
- [Background] Keller A, Leidinger P, Borries A, Wendschlag A, Wucherpfennig F, Scheffler M, Huwer H, Lenhof HP, Meese E. miRNAs in lung cancer - studying complex fingerprints in patient's blood cells by microarray experiments. BMC Cancer. 2009 Oct 6;9:353. doi: 10.1186/1471-2407-9-353. PMID 19807914
- [Background] Leidinger P, Keller A, Meese E. MicroRNAs - Important Molecules in Lung Cancer Research. Front Genet. 2012 Jan 23;2:104. doi: 10.3389/fgene.2011.00104. eCollection 2011. PMID 22303398